CLINICAL TRIAL: NCT01441661
Title: Sunitinib Intake Conditions in the Treatment of Patients With Renal Cell Carcinoma: a Multicenter, Non-interventional, Retrospective Survey
Brief Title: Sunitinib Intake Conditions in the Treatment of Patients With Renal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Cancer Foundation, China (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: CFC20110815
Record Dates: First submitted 2011-09-26; First posted 2011-09-28 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2007-09

CONDITIONS: Renal Cell Carcinoma
Keywords: Sunitinib; kidney diseases; urogenital neoplasms; kidney cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Diseases; Urogenital Neoplasms; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Sunitinib Renal Cell Carcinoma: Patients diagnosed with Renal Cell Carcinoma (RCC) and treated with Sunitinib from 2008 to present will be eligible. This will include current active patients as well as patients who have expired and have medical records available.

SUMMARY:
This non-interventional study includes patients with advanced renal cell carcinoma who are treated with Sunitinib alone or combined with other systemic therapies. The aim of the trial is to increase knowledge about usage, dosage, efficacy and safety under conditions of routine use of Sunitinib.

DETAILED DESCRIPTION:
Because State Food and Drug Administration (SFDA) exempted manufacturers from conducting clinical trials of Sunitinib in China, overall efficacy and safety data of Sunitinib in Chinese patients with renal cell carcinoma were deficiency. The investigators carried out this research project will be sufficient evidence, and help clinicians in China to make decision in real daily practice.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, unresectable advanced renal cell carcinoma;
* Sunitinib as first-line treatment alone or combined with other therapies.

Exclusion Criteria:

* History of Grade 3/4 severe allergic reaction to Sunitinib or its metabolites

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with RCC and treated with Sunitinib from 2008 to present will be eligible. This will include current active patients as well as patients who have expired and have medical records available.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2007-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Disease control rate (DCR) | 2008-2011 (up to 3 years)
  * To determine the Disease control rate (DCR) defined as the percentage of patients who have a partial response (CR) or complete response (PR) to Sunitinib plus those whose disease is stable (DS).
  * To determine the Objective Responsive Rate (ORR) defined as the percentage of patients who have a partial response (PR) or complete response (CR) to Sunitinib.

SECONDARY OUTCOMES:
Progression Free survival (PFS) | 2008 - 2011 (up to 3 years)
  • To assess the Progression Free survival (PFS) as defined by time interval from date of first dose of Sunitinib to date of the progression of cancer or date of death due to any reasons whichever appears earlier.
Overall Survival (OS) | 2008 - 2011 (up to 3 years)
  • To evaluate Overall Survival (OS) as defined by time interval from date of first dose of Sunitinib to date of death due to any reason.
Number of patients with adverse events | 2008 - 2011 (up to 3 years)
  • To evaluate Safety of Sunitinib. Adverse events were graded according to the National Cancer Institute issued the Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Zhangqun Ye, MD, Principal Investigator — Tongji Hospital
Locations (2):
- China (2):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Tongji Hospital, Tongji Medical College of Hust, Wuhan, Hubei